CLINICAL TRIAL: NCT00023101
Title: Lead, Endocrine Disruption and Reproductive Outcomes
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8337-CP-001
Record Dates: First submitted 2001-08-22; First posted 2001-08-24 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Lead Poisoning; Infertility
Keywords: lead; endocrine dysfunction
MeSH Terms: conditions — Lead Poisoning; Infertility

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This prospective cohort study of 400 lead exposed and 400 non-lead exposed women and their husbands assesses endocrine dysfunction and adverse reproductive outcomes. Residing in two study areas in Shenyang, China, the women are married, 20 and 34 years of age, never smokers, have obtained permission to have a child, and have attempted to become pregnant over the course of the study. Lead exposure is defined by lead levels in blood samples collected at the baseline survey (both women and their husbands), first and second trimesters, and at delivery (both maternal and cord blood). Endocrine dysfunction is monitored by urinary hormone metabolites including follicle-stimulating hormone (FSH), luteinizing hormone (LH), estrone conjugates (E1C), and pregnanediol-3-glucuronide (PdG). Reproductive endpoints include menstrual disturbance, time to conception, spontaneous abortion, preterm delivery, and low birth weight.

ELIGIBILITY:
married women who:

* currently reside in two study areas in Shenyang, China
* between 20 and 34 years of age
* never smokers
* have obtained permission to have a child
* are attempting to become pregnant over the course of the study.

Ages: 20 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800
Dates: Start 1996-08